CLINICAL TRIAL: NCT04052269
Title: A Pilot Study to Investigate the Effect of Phosphodiesterase Inhibitors on Chorioretinal Blood Flow Using Optical Coherence Tomography Angiography.
Brief Title: Phosphodiesterase Inhibitors in Glaucoma Study (PhiGS)
Acronym: PhiGS
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: suspended due to COVID
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/WE/5104
Record Dates: First submitted 2019-08-05; First posted 2019-08-09 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Sildenafil Citrate; Tadalafil

STUDY DESIGN:
Intervention Model Description: Healthy vs affected eyes (glaucoma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eyes with glaucoma (Experimental): patients with glaucoma will have imaging of retina post administration of Sildenafil or Tadalafil.
  Interventions: Drug: Sildenafil 100mg
- Healthy (unaffected) eyes (Other): patients with healthy eyes who are already taking Sildenafil or Tadalafil have their imaging of retina post administration of Sildenafil or Tadalafil.
  Interventions: Drug: Sildenafil 100mg

INTERVENTIONS:
Drug: Sildenafil 100mg — study drug (Sildenafil or Tadalafil) administered orally in pill form with glass of water.
  Other Names: Tadalafil

SUMMARY:
It is commonly known that high eye pressure is associated with glaucoma. However, there is also a theory that poor circulation to the eye is a contributing factor. Therefore, if we can increase the flow of blood to the eye, we may be able to stop people losing vision from this disease.

Phosphodiesterase inhibitors (for example sildenafil, tadalafil, Viagra®, Cialis®) are drugs used to improve blood flow to certain parts of the body. They are commonly used on an ad-hoc basis to treat erectile dysfunction, in addition to problems with blood circulation to the lungs, fingers and toes.

The majority of previous work in this field has been completed using insensitive, poorly reproducible techniques such as colour doppler ultrasound. Since then, a new imaging modality able to image blood flow in blood vessels without the need for the injection of contrast has entered clinical use.

This initial pilot study is designed as a proof-of-concept study to investigate whether we can measure detectable changes in the blood flow to the retina and choroid at the back of the eye following ingestion of a phosphodiesterase inhibitor medication by healthy and glaucomatous volunteers already taking this medication for erectile dysfunction.

DETAILED DESCRIPTION:
Hypotheses

This study is examining the hypothesis that Phosphodiesterase inhibitors increase chorio-retinal blood flow; in other words, we hypothesise that drugs like Viagra that have a known effect of generally increasing circulation may also increase the blood flow in the back of the eye -retina, with possible beneficial effect.

Study design

This is a small pilot study which is not expected to produce a definitive answer to our question -however, if successful this study will enable us to progress to a larger study that will have much more data to base our conclusions on.

Our present study will, therefore, examine both healthy and glaucomatous eyes with regards to the level of blood flow in the retina - something that can be measured using optical coherence tomography (OCT), a safe and non-invasive procedure which has been in use as part of the standard of care for some time.

Estimated Timeline

Ethics assessment - April 2019 Patient recruitment - June to Sep 2019 Study period - May 2019 to Jan 2020

Setting

Patient encounters will take place at either the eye clinic, level 1, Charing Cross Hospital, or the iCORG clinical trials unit, Western Eye Hospital.

Encounter 1 - As part of the routine clinic visit potentially eligible patients will be approached by the members of the regular care team and study discussed with those who are interested. Patients who are comfortable to proceed (have discussed the study in detail with the doctor and have had their questions answered satisfactorily)will provide consent which will be documented in writing; those who wish to have more time will be afforded as much time as they need to decide whether or not to participate.

Once the patient has consented to participate, the following study procedures will be done as part of that visit:

Baseline assessment Medical history Baseline assessment Ophthalmic history Baseline assessment Drug history Baseline assessment Allergy history - all of the above will be assessed by the study doctor

Baseline assessment Visual acuity - patient reads letters from a chart 10 feet (3 meters) away to ascertain the quality of vision Baseline assessment Visual field test -non-invasive test where the study doctor examines how much 'side' vision patient has using a computerized machine. Lights are flashed on, and patient has to press a button whenever they see the light.

Baseline assessment Colour vision/contrast sensitivity - patient reads letters /numbers from a multi coloured picture.

Baseline assessment Intraocular pressure (IOP)- Study Doctor places eye drops which numb the eyes and measures the pressure in each eye by gently touching the instrument (called a tonometer) to the front surface of the eye. This is a standard procedure and the numbing eye-drops are safe and have been part of standard care pathway for some time.

Baseline assessment Slit-lamp examination- study doctor examines eyes using a special lens and light Baseline assessment Blood pressure (BP)- standard procedure Baseline assessment OCT and OCTA scan - OCT stands for optical coherence tomography which is a type of imaging technique that is commonly used to image the eye in the clinic, using light to visualise the layers of the back of the eye. There are no risks or discomforts associated with this type of imaging.

Study procedure PDE-5 inhibitor dosing - participants take their drug as per protocol (according to what drug they have been taking) Study procedure OCTA 30 minutes - as OCT but done in different time intervals 30min, 60min, 120min.

Study procedure Repeat BP, IOP at 50 minutes - as described above Study procedure OCTA 60 minutes - as described above Study procedure OCTA 120 minutes- as described above

Upon completion of the study, patients from both cohorts(glaucoma and andrology) will continue their regular care in their usual clinics. The follow-up data routinely generated as part of the glaucoma care pathway (only)which is stored within the hospital data system e.g the central macular thickness, visual fields, IOP and other parameters will be accessed for 3 years following completion of participation with a view of correlating initial results with possible disease progression and other related outcomes. This segment of the study is purely data-based and does not require any active involvement from the patients; participation in the data follow-up part of the study is optional and permission to access the relevant data will be documented in the informed consent form.

Analyses

No interim analyses will take place as they are deemed not needed.

Sampling

Sampling /recruiting for this pilot study will be from consecutive eligible patients from glaucoma and andrology clinics as well as patients recruited via the Western Eye Hospital patient database and replies to poster adverts at Imperial College Healthcare NHS Trust.

The sample size target for this pilot study is 30 including 15 glaucoma subjects and 15 non-glaucoma subjects.

No sample size or power calculations are necessary for this pilot study.

Recruitment sources (aim: 15 non glaucoma participants, 15 glaucoma participants)

Glaucoma clinics (Imperial Healthcare NHS Trust) Andrology clinics (Imperial Healthcare NHS Trust) Western Eye Patient database - potential patients will be contacted by telephone by a member of the usual care team and given the opportunity to receive more information about research that we are undertaking.

Poster (attached) advertisements will be strategically placed in andrology and glaucoma waiting rooms.

They will also have the opportunity to be emailed/posted a patient information sheet and given the opportunity to ask further questions.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent to participate in the study
* Aged between 40 and 80 years of age
* Clear optical media
* Spherical equivalent +-10D
* IOP 21mmHg

Exclusion Criteria:

* have used sildenafil for 48 hours (4 hour half-life) and tadalafil for 5 days (48 hour half-life).
* have a known adverse reaction to any phosphodiesterase inhibitors
* have an inherited photoreceptor disease (manufacturer contra-indication)
* have any other known ocular disease (except glaucoma in this cohort)
* have had non-arteritic anterior ischaemic optic neuropathy (manufacturer precaution due to lack of long term visualfield studies)
* are on current ritonavir, erythromycin, cimetidine treatment (Manufacturer advises if concurrent use of ritonavir is unavoidable, the max. dose should not exceed 25 mg within 48 hours)
* have serious cardiac or liver disease (manufacturer contra-indication)
* have had a stroke or myocardial infarction (manufacturer contra-indication) within 6 months
* have anatomical deformation of the penis or conditions predisposing to priapism (sickle cell anaemia, leukaemia, multiple myeloma)
* have hypotension (manufacturer contra-indication) BP<100/60
* have secondary or narrow/closed angle glaucoma

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Changes in central macular thickness as assessed by retina imaging | 30 minutes, 60 minutes, 120 minutes
  OCT and angiographic findings before and after drug administration including
Changes in retinal vascular density as assessed by retina imaging | 30 minutes, 60 minutes, 120 minutes
  OCT and angiographic findings before and after drug administration including
Changes in outer retina flow as assessed by retina imaging | 30 minutes, 60 minutes, 120 minutes
  OCT and angiographic findings before and after drug administration including
Changes in choroidal vascular density as assessed by retina imaging | 30 minutes, 60 minutes, 120 minutes
  OCT and angiographic findings before and after drug administration including
Changes in central choroidal thickness as assessed by retina imaging | 30 minutes, 60 minutes, 120 minutes
  OCT and angiographic findings before and after drug administration including
Changes in choroidal flow as assessed by retina imaging | 30 minutes, 60 minutes, 120 minutes
  OCT and angiographic findings before and after drug administration including

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Dr Normando, MD, PhD, Principal Investigator — Imperial College London
Locations (1):
- Western Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No